CLINICAL TRIAL: NCT01032044
Title: Confocal Laser Endomicroscopy for Assessment of Neoplasia After Mucosal Ablation or Resection of Gastrointestinal Neoplasia
Brief Title: CLE for Assessment of Neoplasia After Mucosal Ablation or Resection of Gastrointestinal Neoplasia
Acronym: CLEAN-MARGIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mauna Kea Technologies (Industry)
Collaborators: Cellvizio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MKT-2009-BE-01
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Barrett Syndrome; Barrett's Syndrome; Barrett's Esophagus; Barrett Esophagus; Adenocarcinoma
Keywords: Barrett's esophagus; EsoGastroDuodenoscopy; Barrett's carcinoma; adenocarcinoma; Cellvizio; endomicroscopy; probe-based Confocal Laser Endomicroscopy; pCLE; Radio-frequency ablation; Endoscopic mucosal resection; Photodynamic therapy
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard endoscopic evaluation (Active Comparator): Standard high-definition white light endoscopy guided evaluation
  Interventions: Device: Standard endoscopic evaluation
- pCLE-guided evaluation (Experimental): Endoscopic evaluation of BE guided by probe-based Confocal Laser Endomicroscopy (pCLE guided evaluation)
  Interventions: Device: pCLE guided evaluation

INTERVENTIONS:
Device: Standard endoscopic evaluation — Treatment modalities can include endoscopic mucosal resection, radio-frequency ablation or photodynamic therapy
  Arms: Standard endoscopic evaluation
Device: pCLE guided evaluation — Treatment modalities include endoscopic mucosal resection, radio-frequency ablation, or photodynamic therapy. probe-based Confocal Laser Endomicroscopy is used to decide on re-treatment or not, and to guide and evaluate the treatment during the same endoscopic procedure.
  Arms: pCLE-guided evaluation

SUMMARY:
This study focuses on demonstrating the value of probe-based Confocal Laser Endomicroscopy (pCLE) in guiding endoscopic therapeutic procedures in Barrett's Esophagus (BE).

It is a randomized controlled outcomes study including patients already treated for Barrett's Esophagus lesion(s) and undergoing high definition white light endoscopy follow up procedure, with or without pCLE (2 arms will be considered in this study). The procedures will be carried out per standards of practice with appropriately trained physicians.

DETAILED DESCRIPTION:
It is a randomized controlled outcomes study including patients already treated for Barrett's Esophagus lesion(s) and undergoing high definition white light endoscopy follow up procedure, with or without pCLE guided evaluation (2 arms will be considered in this study). The procedures will be carried out per standards of practice with appropriately trained physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BE with Intestinal Metaplasia, Low Grade-IntraEpithelial Neoplasia/High Grade-IntraEpithelial Neoplasia as the original indication for ablative treatment.
* Undergoing any type of endoscopic BE ablation treatment
* <2cm of circumferential BE and <5 total islands of BE on prior to last ablation.
* Age > 18 years
* Ability to provide written, informed consent

Exclusion Criteria:

* Participation in another clinical study
* Circumferential BE
* Complete eradication of BE documented by biopsies
* Inability to obtain biopsies due to anticoagulation, varices, etc.
* Allergy to fluorescein
* Pregnancy
* Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wallace, MD, Principal Investigator — Mayo Clinic Jacksonville, Florida, United States; Anne Osdoit, Study Director — Mauna Kea Technologies, Paris, France
Locations (6):
- United States (4):
  - Mayo Clinic, Jacksonville, Florida
  - University of Chicago Hospital, Chicago, Illinois
  - Veterans Affairs Hospital, Kansas City, Missouri
  - University of Washington Medical Center, Seattle, Washington
- Centre Hospitalier Universitaire, Nantes, France
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Derived] Wallace MB, Crook JE, Saunders M, Lovat L, Coron E, Waxman I, Sharma P, Hwang JH, Banks M, DePreville M, Galmiche JP, Konda V, Diehl NN, Wolfsen HC. Multicenter, randomized, controlled trial of confocal laser endomicroscopy assessment of residual metaplasia after mucosal ablation or resection of GI neoplasia in Barrett's esophagus. Gastrointest Endosc. 2012 Sep;76(3):539-47.e1. doi: 10.1016/j.gie.2012.05.004. Epub 2012 Jun 28. PMID 22749368

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment: Standard high-definition white light endoscopy guided treatment
  Standard endoscopic treatment of BE: Treatment modalities can include endoscopic mucosal resection, radio-frequency ablation or photodynamic therapy
- pCLE-guided Treatment: Endoscopic treatment of BE guided by probe-based Confocal Laser Endomicroscopy
  pCLE guided endoscopic treatment of BE: Treatment modalities include endoscopic mucosal resection, radio-frequency ablation, or photodynamic therapy. probe-based Confocal Laser Endomicroscopy is used to decide on re-treatment or not, and to guide and evaluate the treatment during the same endoscopic procedure.
Period: Overall Study
Arm/Group | Standard Treatment | pCLE-guided Treatment
Started | 82 | 82
Procedure | 74 | 75
Completed | 57 | 62
Not Completed | 25 | 20
Not completed — Protocol Violation | 14 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 11 | 11

BASELINE CHARACTERISTICS:
Population: Exploratory analysis of the data according to the intent-to-treat principle resulted in no suggestion of systematic bias in the two groups regarding withdrawals. Only 1 patient was withdrawn because of intolerance to fluorescein.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Endoscopic Evaluation | pCLE-guided Evaluation | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Continuous [Mean (Full Range); unit: years] | 67.9 [45.4 to 87.2] | 69.6 [50.2 to 86.1] | 68.8 [45.4 to 87.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 78 | 75 | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Barrett's Esophagus (BE) Participants With a Composite Outcome of "Optimally Treated"
Description: Number of Barrett's Esophagus (BE) Participants with a Composite Outcome of "Optimally Treated", in each group defined as patients for whom all lesions are ablated when disease is present, or not ablated when disease is absent, or have complete ablation of all disease at the 3 month follow-up.
Time Frame: 3 month follow-up endoscopic procedure
Population: Among the 141 patients who completed the initial procedure, 119 had follow-up visits.
Measure: Number; unit: participants
Arm/Group | Standard Endoscopic Evaluation | pCLE-guided Evaluation
Number analyzed (Participants) | 57 | 62
participants | 16 | 16

ADVERSE EVENTS:
Time Frame: from inclusion to 3 months follow-up visit post-procedure
Arm/Group | Standard Treatment | pCLE-guided Treatment
Serious Adverse Events (participants affected / at risk) | 0/82 | 1/82
Other Adverse Events (participants affected / at risk) | 0/82 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (N=82) | pCLE-guided Treatment (N=82)
Intolerance to Fluorescein (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No